CLINICAL TRIAL: NCT02705144
Title: Definition of the Status of the Human Lung Stem Cell Niches ex Vivo in Tissue Biopsies Performed in Patients With Emphysema and Interstitial Fibrosis Compared to Non-diseased Areas
Brief Title: Definition of the Status of the Human Lung Stem Cell Niches ex Vivo in Tissue Biopsies Performed in Patients With Emphysema and Interstitial Fibrosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Weizmann Institute of Science (Other)
Responsible Party: Principal Investigator, Dr. Tiberiu Shulimzon MD, Director Interventional Pulmonology Unit, Sheba Medical Center
Other Study IDs: SMC -15 - 2787
Record Dates: First submitted 2016-02-21; First posted 2016-03-10 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Lung Diseases, Interstitial
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Lung tissue biopsies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- biopsies from lung tissue affected by emphysema: analysis of the number of stem cell niches
  Interventions: Other: analysis of the number of stem cell niches
- biopsies from lung tissue affected by interstitial fibrosis: analysis of the number of stem cell niches
  Interventions: Other: analysis of the number of stem cell niches
- biopsies from normal appearance lung tissue: analysis of the number of stem cell niches
  Interventions: Other: analysis of the number of stem cell niches

INTERVENTIONS:
Other: analysis of the number of stem cell niches — to assess stem cell compartments in their niches and their proliferative and developmental properties in vitro

SUMMARY:
To characterize stem cell compartments in their niches in different clinical situations (non-diseased compared to emphysematous and fibrotic pulmonary tissue) and to assess their proliferative and developmental properties in vitro.

To further implement lung organoid culture system in the drug screening and development of patient personalized medicine.

DETAILED DESCRIPTION:
Scientific Background

Degenerative lung disorders are the result of inflammatory events that end in destruction of the normal pulmonary architecture. Two main patterns exist:

1. Chronic obstructive lung disease (COPD) is a major cause of morbidity and mortality. Until 2020 it is expected to become the third cause of mortality following cardiovascular disorders and cancer. Emphysema is the destructive form of COPD as the alveolated tissue disappears. This anatomic pattern is not always homogenous and functional impairment is not connected to the extent of the tissue destruction. Therapeutic elimination of the destroyed tissue may be achieved by surgery or by using various blocking techniques (Lung Volume Reduction).
2. Pulmonary fibrosis (PF) is characterized by abnormal repair of the respiratory epithelium. Various diseases may result in PF such as infections, autoimmune (connective tissue disorders), sarcoidosis, hypersensitivity pneumonitis, pneumoconiosis, histiocytosis X, lymphangioleiomyomatosis LAM etc. In many situations a cause effect relationship cannot be identified and the disease is idiopathic IPF.

During the last years cell based therapies using progenitor cells and various scaffolds became available in various medical fields. Lung regenerative medicine appears to be an alternative to transplantation in these end-stage diseases.

However, very complex cellular composition of the lung, comprising more than 40 different cell types, makes this objective challenging. The epithelial lining of the respiratory tract, composed of conducting and respiratory parts, varies along its proximo-distal axis. The conducting airways from the trachea to bronchioles of human lungs consist of pseudostratified epithelium, comprising equal proportions of basal cells, secretory cells, and ciliated cells, as well as some neuroendocrine cells. The smallest bronchioles, known as terminal and respiratory bronchioles, are lined with a simple columnar or cuboidal epithelium containing secretory and ciliated cells with fewer basal cells. The epithelia of these conducting airways form a tight barrier against the outside world and are specialized for the process of mucociliary clearance. The alveoli are lined by type 1 and 2 alveolar epithelial cells, called AT1 and AT2, respectively, hereafter. These cells are also specialized for barrier function and the extremely thin AEC1s share a basement membrane with the surrounding network of pulmonary capillaries to facilitate the diffusion of gases between the atmosphere and the circulation.

This general distribution of epithelial cell types is conserved between humans and model organisms such as rodents. However, there are notable differences. For example, the transition from a pseudostratified to columnar epithelium occurs more proximally in rodents, so only the trachea and mainstem bronchi are lined with a pseudostratified epithelium. Nearly all intralobar airways in mice are lined with a simple columnar or cuboidal epithelium with few basal cells. In mice, the abrupt transition from a conducting airway to the alveoli is known as a broncho-alveolar duct junction. In humans, terminal bronchioles give rise to respiratory bronchioles from which many alveolar ducts terminate ultimately in alveoli. Considering essential role of epithelial compartment in the lung much effort has been done to identify epithelial stem and progenitor cells responsible for regenerative and reparative functions.

Epithelial progenitors reside in unique microenvironment or niches, represented by vascular and mesenchymal cells, which are richly innervated. This architecture highly resembles HSM niches.

Considerable progress has been made in mice toward identifying the signals that regulate lung epithelial stem cell self-renewal and differentiation. These include Notch, Hippo/Yap, ROS/Nrf2, EGF, FGF, c-myb, and cytokines including IL-4, -13 and -6. Neighboring epithelial cells, stromal cells (including mesenchymal cells, fibroblasts, smooth muscle cells, and endothelium) and immune cells all represent potential sources for these factors. Distinct stem cell niches have been defined in adult mouse trachea and lung in the steady state and there is increasing evidence that in different pathological conditions stem cell niches are affected and altered.

Very little is known about stem cells and stem cell niches in human adult lung and the signals which regulate maintenance of the lung tissue homeostasis in health and disease.

Recently, the Reisner group at the Weizmann Institute has demonstrated that vacating the lung stem cell niches is a pre-requisite for successful transplantation of mouse or human lung progenitors (Nature Medicine 2015). To that end, they used an initial lung injury with naphthalene which triggered an immediate stimulation of endogenous progenitors. Thus within 48 hours the dividing progenitors could be effectively ablated by 6 Gy total body irradiation enabling effective engraftment of donor lung progenitors (Fig.1).

Fig. 1: Engraftment and functional repair of injured lungs by mouse embryonic lung cells. Following lung injury with NA and conditioning with 6Gy TBI, C57BL/6 adult mice were transplanted with syngeneic E16 stage embryonic lung cells from GFP+ donors. (a,b) Representative two-photon microscopy extended focus images of the lungs of transplanted mice 6 weeks after transplantation, showing entire scan depth from top to bottom of chimeric lung, without (a: z-stack 88μm), and with (b) co-staining of blood vessels with Quantum dots (red) (bar=90μm). (c) Two-photon extended focus image, showing entire scan depth from top to bottom of chimeric lung (z-stack 96μm) 16 weeks post-transplantation. (d) Two-photon microscopy of non-transplanted C57BL mouse lung showing background (bar=90μm). (e,f,g) Representative images of chimeric lungs stained with anti-GFP (green) and anti-AQP-5 (red), indicating incorporation of donor-derived type I alveocytes into the gas-exchange surface. (h,i,j) Chimeric lung stained with anti-GFP (green), anti-Sp-C antibodies (blue), demonstrating donor-derived surfactant producing type II alveocytes (bars=20μm). All the individual images shown above are representative of n=10 mice pooled from 3 independent experiments. (m,n) Lung function measurements 6 weeks after transplantation. (k,l) Staining of chimeric lung for CFTR (red) and (GFP), demonstrating CFTR positive donor cells. (m) Lung baseline compliance. Comparison of control intact mice vs mice with lung injury (Student's t-test, P<0.001), and of mice with lung injury vs mice transplanted after injury (Student's t-test, P=0.008). (n) Tissue damping. Comparison of control mice vs mice with lung injury (Student's t-test, P=0.015), and of mice with lung injury vs mice transplanted after injury (Student's t-test, P=0.021). Values are means ± SEM of 10-15 (n=15 control, n=10 injured and n=10 treated) mice in each group pooled from two independent experiments However, while this conditioning was required for enabling effective engraftment of donor lung progenitors in normal mice, we envision that in patients with different lung diseases, the lung niches could be already partially depleted and therefore transplantation might require less severe conditioning.

Objective To characterize stem cell compartments in their niches in different clinical situations (non-diseased compared to emphysematous and fibrotic pulmonary tissue) and to assess their proliferative and developmental properties in vitro.

To further implement lung organoid culture system in the drug screening and development of patient personalized medicine.

Methods Biopsies of lung tissue will be obtained by surgical procedures: open lung biopsies. This procedure is routinely performed for histological diagnosis of fibrotic diseases. Patients with emphysema and end stage fibrotic disease are at higher risk to develop lung cancer. A large proportion of surgically treated lung cancer patients have emphysema and fibrotic disease as histologic background. Lobectomy and pneumonectomy are frequently performed as state of the art procedures in lung cancer surgical management. Part of the resected lung tissue contain emphysematous and fibrotic changes or make look macroscopically and microscopically normal. These "non-cancerous" areas will be sampled and preserved at the Sheba Tissue Bank for evaluation together with samples from fibrotic and emphysematous areas. The biopsies will be analyzed by immunohistology, FACS and 3D organoids (after the removal of fibroblasts) at the immunology laboratory at Weizmann Institute.

All Samples will be collected following informed consent signatures of patients both on the designated informed consent form for this protocol and the tissue bank form. We may have as many as 3-4 patients/ week. Collected samples will be resected by experienced personnel either from the Thoracic Surgery Department or the Pathology Department (as part of their job description in the Tissue Bank). Fresh samples will be transported to the Weizmann institute for FACS and IHC.

As very limited knowledge exists on human lung tissues it will be mandatory to test lung tissues from healthy and diseased lungs. Initially we suggest testing 10-15 normal lung tissues and 15-20 diseased samples during the period of 2 years. As mentioned before the normal lung tissues will be obtained as "non-cancerous" areas from patients undergoing lobectomies/pneumonectomies.

ELIGIBILITY:
Inclusion Criteria:

* lung emphysema, lung interstitial fibrosis, lung cancer patients

Exclusion Criteria:

* lung infectious diseases (bronchiectasis, lung abscess, pneumonia)
* pulmonary edema

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lung emphysema and interstitial lung disease as the background for lung cancer
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
The number of stem cell compartments in their niches in different clinical situations (non-diseased compared to emphysematous and fibrotic pulmonary tissue) . | 2 years

SECONDARY OUTCOMES:
The number of organoids in their cellular positions | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosen C, Shezen E, Aronovich A, Klionsky YZ, Yaakov Y, Assayag M, Biton IE, Tal O, Shakhar G, Ben-Hur H, Shneider D, Vaknin Z, Sadan O, Evron S, Freud E, Shoseyov D, Wilschanski M, Berkman N, Fibbe WE, Hagin D, Hillel-Karniel C, Krentsis IM, Bachar-Lustig E, Reisner Y. Preconditioning allows engraftment of mouse and human embryonic lung cells, enabling lung repair in mice. Nat Med. 2015 Aug;21(8):869-79. doi: 10.1038/nm.3889. Epub 2015 Jul 13. PMID 26168294
- [Background] Raghu G, Rochwerg B, Zhang Y, Garcia CA, Azuma A, Behr J, Brozek JL, Collard HR, Cunningham W, Homma S, Johkoh T, Martinez FJ, Myers J, Protzko SL, Richeldi L, Rind D, Selman M, Theodore A, Wells AU, Hoogsteden H, Schunemann HJ; American Thoracic Society; European Respiratory society; Japanese Respiratory Society; Latin American Thoracic Association. An Official ATS/ERS/JRS/ALAT Clinical Practice Guideline: Treatment of Idiopathic Pulmonary Fibrosis. An Update of the 2011 Clinical Practice Guideline. Am J Respir Crit Care Med. 2015 Jul 15;192(2):e3-19. doi: 10.1164/rccm.201506-1063ST. PMID 26177183
- [Background] Sanchez-Salcedo P, Wilson DO, de-Torres JP, Weissfeld JL, Berto J, Campo A, Alcaide AB, Pueyo J, Bastarrika G, Seijo LM, Pajares MJ, Pio R, Montuenga LM, Zulueta JJ. Improving selection criteria for lung cancer screening. The potential role of emphysema. Am J Respir Crit Care Med. 2015 Apr 15;191(8):924-31. doi: 10.1164/rccm.201410-1848OC. PMID 25668622